CLINICAL TRIAL: NCT04060238
Title: Investigation of the Effect of Protanopia ("Red Blindness") on the Brightness Perception of Brake Lights and Their Effect on Reaction Time
Brief Title: Effect of Protanopia on the Brightness Perception of Brake Lights
Acronym: ProLight
Status: Completed | Type: Observational
Sponsor: Aalen University (Other)
Collaborators: Karlsruhe Institute of Technology (KIT), Karlsruhe/FRG (Unknown)
Responsible Party: Sponsor
Other Study IDs: ProLight_I
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2019-06

CONDITIONS: Color Blindness, Red; Reaction Time
Keywords: protanopia; taillight; brake light; differential luminance sensitivity; contrast sensitivity; colour vision; colour vision defect; perimetry; semi-automated kinetic perimetry; traffic; motorist; reaction time
MeSH Terms: conditions — Color Vision Defects

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal colour vision: Normal trichromopsia
  Interventions: Diagnostic Test: Anomaloscope (colour vision test)
- Inherited red blindness: Protanopia
  Interventions: Diagnostic Test: Anomaloscope (colour vision test)

INTERVENTIONS:
Diagnostic Test: Anomaloscope (colour vision test) — The Heidelberg Multi Colour (HMC) Anolmaloscope (Oculus Inc., Dutenhofen/FRG) is used to differentiate between normal controls (normal trichromatopsia) and test subjects with protanopia ("inherited red colour blindness")

SUMMARY:
The aim of the offered project is to investigate the influence of protanopia (red blindness) or protanomaly (red vision weakness) on the recognizability of red brake lights with the help of a test person study. From this, estimates of the influence of protanopia or protanomaly on driving ability are to be derived.

If a relevant influence can be demonstrated in the study, recommendations for action for the legislator will be made.

Translated with www.DeepL.com/Translator

DETAILED DESCRIPTION:
Protanopia is an x-chromosomal inherited cone pigment disorder that related to the red cone,i.e. the L-cone function completely fails. The prevalence of protanopia in the male population is 1%. An incomplete impairment of the L-cone is called protanomaly. The prevalence here is also in 1% of the male population.

In comparison to persons with normal vision red objects appear darker for persons with missing or functionally limited L-cones. This is particularly critical in road traffic, where red is used as a signal colour, for example in traffic lights or brake lights is used.

The scientific questions that need to be investigated are as follows:

1. At which contrast threshold (relative brightness) does a proband with protanopia recognize a brake light compared to a normal person?
2. If the luminance determined is above the contrast threshold, what influence does the excess of the contrast or the determined luminance have on the reaction time?
3. Are there differences with regard to the technology used in the brake light (incandescent lamp or LED)?

For this purpose, a representative set of combination rear lamps, focusing on stoplight, taillight (and of the elevated brake light) in a static situation is created. The test setup is based on a driving pursuit scenario. The test person is positioned at a relevant distance to the combination of rear lamps.

To determine the threshold contrast, an algorithm is developed to control the relative brightness of the brake lights and integrated into the test sequence control. In addition, a method for automated determining of the related reaction time is implemented.

Two taillight technologies (incandescent lamp and LED) are examined at both ambient brightness levels: (i) "bright", i.e. photopic luminance level (Lu >> 10 cd/m2) and (ii) "dark", i.e. mesopic luminance level (Lu < 10 cd/m2).

A comprehensive ophthalmological/optical examination (including visual acuity, ocular alignment, ocular motility, assessment of the leading eye, testing of the efferent and afferent pupillary system and biomicroscopic inspection of the anterior and posterior segments of the eye) is carried out. Comprehensive colour vision testing it performed with the HMC anomaloscope, Oculus Inc., Dutenhofen/FRG, including assessment of the loss of brightness sensation during anomaloscopic exam with max. red. stimulus . In addition, standardized semi-automated kinetic perimetry (SKP) along the horizontal meridian with an automated perimeter (Octopus 900, Haag-Streit Inc., Koeniz/CH) is performed. The ratio of the horizontal extent ("diameter") obtained with both, red vs. white stimuli, is measured and taken as a clinical parameter for quantifying the magnitude of the individual "protan colour vision deficiency".

To illustrate the worst-case scenario, this study is limited to protanopic patients. It is intended as a pure comparative study between a "protanopic" patient group and a "normal vision" control group. The protanopic test subjects and the control subjects are matched with regard to gender and age.

This study is carried out in a "within-subject design", i.e. all test persons go through all situations. In order to minimize sequence effects, the related test conditions are randomized.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* male
* age (greater or equal) 18 years

Exclusion Criteria:

* binocular (high contrast) distant visual acuity worse than 0.8 (16/20)
* spherical ametropia exceeding 8 dpt
* cylindrical ametropia exceeding 2.5 dpt
* manifest strabismus (squint) with diplopia
* relative afferent pupillary defect exceeding 0.3 log units
* anamnestic (patient history) OR morphological (slit lamp --> anterior segment, ophthalmoscope --> retina) clue/indicator for a ophthalmologically relevant affection of the eye OR the visual pathway
* S.p. severe ocular trauma
* Current OR s.p. severe intraocular inflammation
* S.p. intraocular surgery within the past three months

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — male subjects only
Study Population: Ophthalmologically normal (male) subjects OR (male) subjects with (inherited) protanopia (red blindness)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity (I) | within one year
  Contrast sensitivity between taillight and brake light under two luminance conditions

SECONDARY OUTCOMES:
Reaction time | within one year
  Time span within the onset of the brake light and the reaction of the tested subject
Contrast sensitivity (II) | within one year
  taillight technology: incandescent lamp vs. light emitting diode (LED)
Reaction time (II) | within one year
  taillight technology: incandescent lamp vs. light emitting diode (LED)
Perimetric extent of horizontal meridian | within one year
  (Semi-autmated kinetic) perimetry with white vs. red stimuli
Loss of brightness sensation during anomaloscopic exam | within one year
  Loss of brightness sensation during anomaloscopic exam with max. red. stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, MD, Study Chair — Aalen University of Applied Sciences
Locations (1):
- Ulrich SCHIEFER, Aalen, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: Undecided
In case of a subsequent study, aiming at assessing the colour sensitivity of single cones, pseudonomized participant data will be shared with the involved researchers.